CLINICAL TRIAL: NCT05401422
Title: Efficacy and Safety of Combining Doxycycline With Pulsed Dye Laser Versus Topical Brimonidine 0.33% in the Treatment of Erythematotelangiectatic Rosacea: a Comparative Clinical and Dermoscopic Study
Brief Title: Brimonidine in Rosacea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rosacea
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulsed dye laser (Active Comparator): Laser
  Interventions: Other: treatment
- Doxycycline (Active Comparator): Drug
  Interventions: Other: treatment
- Brimonidine gel 0.33% (Active Comparator): Topical drug
  Interventions: Other: treatment

INTERVENTIONS:
Other: treatment — types

SUMMARY:
Rosacea is a chronic and relapsing inflammatory cutaneous disorder with highly variable prevalence worldwide.

DETAILED DESCRIPTION:
In our study, we will compare the safety, efficacy, and adverse effects of low-dose oral doxycycline alone versus combined with pulsed dye laser or topical brimonidine in treating erythematotelangiectatic rosacea in an attempt to build a treatment strategy in a disease with complex pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with current erythematotelangiectatic rosacea

Exclusion Criteria:

- Pregnant females. 2-Patients on systemic steroids. 3-Patients complaining of other dermatological disorders mainly photosensitive cutaneous disorder.

4- Patients receiving any systemic treatment including retinoids for the previous 1 month or any topical treatment for the previous 2 weeks or any laser sessions for the previous 3months for erythematotelangiectatic rosacea at least.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-05-25 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical erythema assessment scale | 3 months
  clinical scale

SECONDARY OUTCOMES:
Thickness of capillaries by dermoscope | 3 months
  Assessment